CLINICAL TRIAL: NCT03255473
Title: High Dose Oral Steroids in Sudden Sensorineural Hearing Loss
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: On hold due to COVID-19 outbreak
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-2342
Record Dates: First submitted 2017-08-16; First posted 2017-08-21 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Sudden Sensorineural Hearing Loss (SSNHL)
MeSH Terms: conditions — Hearing Loss, Sudden | interventions — Dexamethasone; dexamethasone 21-phosphate; Prednisone

STUDY DESIGN:
Intervention Model Description: Compare hearing outcomes between treatment with dexamethasone versus prednisone in participants who have been diagnosed with unilateral SSNHL within six weeks, and compare side effect profiles between the two treatment regimens of either dexamethasone or prednisone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone (Active Comparator): All subject identification (ID) numbers will be randomly assigned to the dexamethasone or the prednisone arm of the trial prior to the initiation of the study.
  Interventions: Drug: Dexamethasone
- Prednisone (Active Comparator): All subject ID numbers will be randomly assigned to the dexamethasone or the prednisone arm of the trial prior to the initiation of the study.
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Dexamethasone — All subject ID numbers will be randomly assigned to the dexamethasone or the prednisone arm of the trial prior to the initiation of the study.
  Other Names: dexamethasone sodium phosphate
  Arms: Dexamethasone
Drug: Prednisone — All subject ID numbers will be randomly assigned to the dexamethasone or the prednisone arm of the trial prior to the initiation of the study.
  Other Names: Deltasone
  Arms: Prednisone

SUMMARY:
Compare hearing outcomes between treatment with dexamethasone versus prednisone in participants who have been diagnosed with unilateral SSNHL (sudden sensorineural hearing loss).

DETAILED DESCRIPTION:
Sudden sensorineural hearing loss (SSNHL) affects approximately 5 to 20 per 100,000 persons with spontaneous recovery seen in 32% to 65%. Many different treatments have been investigated in attempt to improve hearing outcomes, with oral corticosteroids having some success. Steroid regimens are highly variable, however, retrospective data has suggested greater improvement in hearing outcomes with the use of high dose oral steroids (dexamethasone) in the setting of unilateral sudden sensorineural hearing loss compared to traditional medical therapy with lower dose oral prednisone. The investigators hypothesize that patients with unilateral SSNHL who are randomized to treatment with high doses of oral dexamethasone will show better hearing outcomes than patients who are randomized to the more common standard clinical practice treatment with lower doses of oral prednisone.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 80 years old
* Present to the Otology or Otolaryngology Clinic at the University of Colorado Hospital with unilateral sudden sensorineural hearing loss (SSNHL)
* Seen within six weeks of initial hearing loss
* Unilateral hearing loss at screening as defined by:

  * Loss of 30 decibels (dB) HL or greater over 3 continuous frequencies with participants reporting that this hearing loss occurred within 3 days
* Present with primary complaint of sensorineural hearing loss
* Normal tympanometry (Type A)
* Normal tympanic membrane

Exclusion Criteria:

* Participants for whom high dose corticosteroids are a contraindicated due to:

  * Pregnancy
  * Known allergies to corticosteroids
  * Other concurrent medical conditions and or medications where high dose oral corticosteroids are not safe to use
* Participants who have Type 1 or Type 2 diabetes
* Participants who have previously received a course of oral steroids for this indication
* Participants who have bilateral SSNHL
* Participants with conductive hearing loss, mixed hearing loss (sensorineural and conductive), or any type of hearing loss that is not SSNHL (i.e. caused by acoustic or physical trauma to the ear)
* Participants with the following conditions/situations will be excluded because the possibility that these could cause SSNHL:

  * History of previous/recurrent unilateral SSNHL
  * History of fluctuating hearing in either ear
  * History of Meniere's syndrome
  * History of chronic granulomatous or suppurative otitis media or cholesteatoma in either ear
  * History of otosclerosis in either ear
* Participants with the following conditions/situations will be excluded due to risk of misclassification of diagnosis of idiopathic SSNHL or because these participants are at higher risk for potential steroid side effects due to other comorbidities. If the time line is not otherwise stated, then the participant will be excluded if they experienced these criteria at any point in their lifetime:

  * Received oral steroids (for any indication besides SSNHL) for greater than 21 days in the preceding 30 days
  * Systemic fungal infections in the last 6 months
  * History of tuberculosis or history of prophylactic tuberculosis treatment for positive skin test (PPD)
  * History of unstable angina, coronary artery stenting or bypass graft within 3 months
  * History of transient ischemic attacks, cardiac arrhythmia, or stroke in the last 4 weeks
  * Serious psychiatric disease or history of psychiatric reaction to corticosteroids, specifically bipolar, schizophrenia, episodes of mania or delirium
  * Prior treatment with chemotherapy agents, immunosuppressive drugs, cyclosporine, or interferon
  * Pancreatitis in the last year
  * Active peptic ulcer disease or history of gastrointestinal bleeding in the last year
  * History of known HIV, hepatitis C, or hepatitis B infection
  * Chronic renal insufficiency requiring dialysis
  * Active shingles (herpes zoster infection)
  * Advanced/severe osteoporosis or nonsurgical aseptic necrosis of the hip

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Changes in Hearing Threshold (Hearing Improvement) | Baseline, 1 week, 1 month, 3 months
  Pure tone averages (from pure tone audiometry) will be recorded for participants at each visit, and assessed for changes in pure tone average over time. Based on a change in pure tone average, participants will be categorized into the different groups.

SECONDARY OUTCOMES:
Changes in Word Recognition Scores | 1 week, 1 month, 3 months, and assessed for change from baseline score.
  Word recognition scores from speech audiometry tests will be summarized, by treatment arm, as a continuous variable using the mean, standard deviation, median, 25th percentile, 75th percentile, minimum and maximum.
Changes in Pure Tone Averages | 1 week, 1 month, 3 months, and assessed for change from baseline pure tone average..
  Continuous pure tone averages calculated from pure tone audiometry will be summarized using the mean, standard deviation, median, 25th percentile, 75th percentile, minimum and maximum and will be presented by treatment arm.
Clinical Frequency Analysis Based on Hearing Improvement | Baseline, 1 week, 1 month, 3 months
  The frequency of patients presenting in each clinical category of hearing improvement will be presented by treatment arm. Hypothesis testing will be performed, using a Mantel-Haenszel Chi-Square test, to test for the association between treatment group and the ordered levels of clinical category of hearing improvement.
Clinical Percentage Analysis Based on Hearing Improvement | Baseline, 1 week, 1 month, 3 months
  The percentage of patients presenting in each clinical category of hearing improvement will be presented by treatment arm. Hypothesis testing will be performed, using a Mantel-Haenszel Chi-Square test, to test for the association between treatment group and the ordered levels of clinical category of hearing improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P Cass, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No